CLINICAL TRIAL: NCT02908620
Title: A Double-blind, Partial Cross-over, Incomplete Factorial Study to Assess the Local Anesthetic Efficacy and Safety of CTY-5339 Anesthetic Spray (CTY-5339-A) When Applied to the Cheek Mucosal Tissue in Normal Volunteers
Brief Title: Experimental Pain Study to Assess Local Anesthetic Efficacy and Safety of CTY-5339 Anesthetic Spray in Normal Volunteers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cetylite Industries (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: C-002
Record Dates: First submitted 2016-09-02; First posted 2016-09-21 (Estimated); Results first posted 2019-07-02 (Actual); Last update posted 2019-07-02 (Actual); Status verified 2019-06

CONDITIONS: Anesthesia
MeSH Terms: interventions — Benzocaine; Tetracaine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (4):
- One spray CTY-5339-A, then one spray CTY-5339-CB (Experimental): A single spray of CTY-5339-A Anesthetic Spray (14.0% benzocaine and 2.0% tetracaine HCl) tested over a 60 minute session, followed by a 4-14 day washout period, followed by a single spray of CTY-5339-CB Anesthetic Spray (14.0% benzocaine) tested over a 60 minute session.
  Interventions: Combination Product: One spray CTY-5339-A; Drug: One spray CTY-5339-CB
- 2 sprays CTY-5339-A, then 1 spray CTY-5339-CB +1 spray placebo (Experimental): Two sprays of CTY-5339-A Anesthetic Spray (14.0% benzocaine and 2.0% tetracaine HCl) tested over a 60 minute session, followed by a 4-14 day washout period, followed by a single spray of CTY-5339-CB Anesthetic Spray (14.0% benzocaine) and a single spray of vehicle control (CTY-5339-P) (sprayed outside the circumscribed area to avoid dilution of active drug) tested over a 60 minute session.
  Interventions: Combination Product: Two sprays CTY-5339-A; Drug: One spray CTY-5339-CB in combination with one spray CTY-5339-P (vehicle control: placebo)
- One spray of CTY-5339-CB, then one spray CTY-5339-A (Experimental): A single spray of CTY-5339-CB Anesthetic Spray (14.0% benzocaine) tested over a 60 minute session, followed by a 4-14 day washout period, followed by a single spray of CTY-5339-A Anesthetic Spray (14.0% benzocaine and 2.0% tetracaine HCl) tested over a 60 minute session.
  Interventions: Combination Product: One spray CTY-5339-A; Drug: One spray CTY-5339-CB
- 1 spray CTY-5339-CB +1 spray placebo, then 2 sprays CTY-5339-A (Experimental): A single spray of CTY-5339-CB Anesthetic Spray (14.0% benzocaine) and a single spray of vehicle control (CTY-5339-P) (sprayed outside the circumscribed area to avoid dilution of active drug) tested over a 60 minute session, followed by a 4-14 day washout period, followed by a two sprays of CTY-5339-A Anesthetic Spray (14.0% benzocaine and 2.0% tetracaine HCl) tested over a 60 minute session.
  Interventions: Combination Product: Two sprays CTY-5339-A; Drug: One spray CTY-5339-CB in combination with one spray CTY-5339-P (vehicle control: placebo)

INTERVENTIONS:
Combination Product: One spray CTY-5339-A — Metered spray bottle with ≈200 uL total spray volume. Contains the active ingredients: 14.0% Benzocaine (USP = 28 mg) and 2.0% Tetracaine Hydrochloride (USP = 4 mg). Administered in a single anesthetic spray.
  Other Names: CTY-5339-A; CTY-5339 Anesthetic Spray; benzocaine; tetracaine; tetracaine HCl; 14.0% benzocaine; 2.0% tetracaine HCl; 2.0% tetracaine; 14.0% benzocaine and 2.0% tetracaine HCl; 14.0% benzocaine and 2.0% tetracaine; benzocaine and tetracaine HCl; benzocaine and tetracaine
  Arms: One spray CTY-5339-A, then one spray CTY-5339-CB; One spray of CTY-5339-CB, then one spray CTY-5339-A
Drug: One spray CTY-5339-CB — Metered spray bottle with ≈200 uL total spray volume. Contains the active ingredient: 14.0% Benzocaine (USP = 28 mg). Administered in a single anesthetic spray.
  Other Names: CTY-5339-CB; benzocaine; 14.0% benzocaine
  Arms: One spray CTY-5339-A, then one spray CTY-5339-CB; One spray of CTY-5339-CB, then one spray CTY-5339-A
Combination Product: Two sprays CTY-5339-A — Metered spray bottle with ≈400 uL total spray volume. Contains the active ingredients: 14.0% Benzocaine (USP = 56 mg total) and 2.0% Tetracaine Hydrochloride (USP = 8 mg total). Administered in two anesthetic sprays.
  Other Names: CTY-5339-A; CTY-5339 Anesthetic Spray; benzocaine; tetracaine; tetracaine HCl; 14.0% benzocaine; 2.0% tetracaine HCl; 2.0% tetracaine; 14.0% benzocaine and 2.0% tetracaine HCl; 14.0% benzocaine and 2.0% tetracaine; benzocaine and tetracaine HCl; benzocaine and tetracaine
  Arms: 1 spray CTY-5339-CB +1 spray placebo, then 2 sprays CTY-5339-A; 2 sprays CTY-5339-A, then 1 spray CTY-5339-CB +1 spray placebo
Drug: One spray CTY-5339-CB in combination with one spray CTY-5339-P (vehicle control: placebo) — A single spray of CTY-5339-CB in a metered spray bottle with ≈200 uL total spray volume, containing the active ingredient: 14.0% Benzocaine (USP = 28 mg). This was administered in combination with a single spray of CTY-5339-P (acting as vehicle control placebo with no active ingredient) in a metered spray bottle with ≈200 uL total spray volume. This combination was used to maintain double-blind conditions. The vehicle control was sprayed outside the circumscribed area to avoid dilution of active drug.
  Other Names: CTY-5339-CB and Placebo; CTY-5339-CB and Vehicle Control; CTY-5339-CB and Control; benzocaine; benzocaine and Placebo; benzocaine and Vehicle Control; benzocaine and Control; 14.0% benzocaine; 14.0% benzocaine and Placebo; 14.0% benzocaine and Vehicle Control; 14.0% benzocaine and Control
  Arms: 1 spray CTY-5339-CB +1 spray placebo, then 2 sprays CTY-5339-A; 2 sprays CTY-5339-A, then 1 spray CTY-5339-CB +1 spray placebo

SUMMARY:
The purpose of this study is to determine if the topical application to cheek tissue of the combination of benzocaine and tetracaine has a longer duration of local anesthetic activity than benzocaine alone.

DETAILED DESCRIPTION:
In a blinded study, either benzocaine alone of the combination of benzocaine and tetracaine will be sprayed onto the cheek mucosal tissue. Onset and duration of local anesthesia will be evaluated over a one hour period using pin prick and QST heat stimulation. Subjects will receive both treatments in a cross-over design with each session separated by 5-7 days. A total of 76 subjects (normal volunteers) will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects between 18-75 years of age with a Body Mass Index (BMI) ≤32;
* Subjects are ASA Category I or II and are in normal physical health as judged by physical and laboratory examinations;
* Subjects with normal appearance of the oral mucosal tissues;
* Subjects must agree to refrain from ingesting any systemic or topical analgesic medication for 3 days or 5 half-lives of the drug prior to and during the study period and alcohol for 1 day prior to and during the study period;
* Subjects must agree to refrain from using mouth rinses, cough drops or throat lozenges on the day of each test session;
* Female subjects must be physically incapable of childbearing potential (postmenopausal for more than 1 year or surgically sterile) or practicing an acceptable method of contraception (hormonal, barrier with spermicide, intrauterine device, vasectomized or same sex partner, or abstinence). Subjects using hormonal birth control must have been on a stable dose of treatment for at least 30 days and received at least 1 cycle of treatment prior to randomization. At Screening and at Baseline of both sessions, all females of childbearing potential must have a negative urine pregnancy test and not be breastfeeding;
* Negative urine drug screen for drugs of abuse at Screening and at Baseline for each Study Session. A positive drug screen result may be permitted if the subject has been on a stable dose of an allowed medication for >30 days;
* The subject is capable of reading, comprehending, and signing the informed consent form.

Exclusion Criteria:

* Subjects with a history of any significant hepatic, renal, endocrine, cardiac, neurological, psychiatric, gastrointestinal, pulmonary, hematologic, or metabolic disorders, including glaucoma, diabetes, emphysema, and chronic bronchitis;
* Subjects with a history of any type of cancer other than skin related cancers;
* Subjects with conditions that affect the absorption, metabolism, or passage of drugs out of the body, (e.g., sprue, celiac disease, Crohn's disease, colitis, or liver, kidney, or thyroid conditions);
* Subjects with any history of alcohol or substance abuse (including a positive drug screen test);
* Subjects that currently have or have a history of uncontrolled hypertension;
* Subjects with a known hypersensitivity to any local anesthetic drug;
* Subjects with a hematocrit level significantly below the normal range on the screening laboratory examination (as judged by the PI);
* Subjects with any clinically significant abnormal lab result (as judged by the PI);
* Subjects with any condition or history felt by the Investigator to place the subject at increased risk;
* Subjects who have smoked or chewed tobacco-containing substances within 6 months prior to the start of the study;
* Subjects judged by the Investigator to be unable or unwilling to comply with the requirements of the protocol;
* Subjects who have used an investigational drug within 30 days prior to entering the study;
* Subjects who have donated blood within 3 months prior to the start of the study;
* Subjects who have previously participated in the trial;
* Subjects who are members of the study site staff directly involved with the study or a relative of the Sponsor or other personnel involved with the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-12-07 (Actual); Primary Completion 2017-04-02 (Actual); Study Completion 2017-06-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elliot V Hersh, DMD, Ph.D., Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, School of Dental Medicine Department of Oral & Maxillofacial Surgery, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang S, Giannakopoulos H, Lowstetter J, Kaye L, Lee C, Secreto S, Ho V, Hutcheson MC, Farrar JT, Wang P, Doyle G, Cooper SA, Hersh EV. Lack of Methemoglobin Elevations After Topical Applications of Benzocaine Alone or Benzocaine Plus Tetracaine to the Oral Mucosa. Clin Ther. 2017 Oct;39(10):2103-2108. doi: 10.1016/j.clinthera.2017.08.017. Epub 2017 Sep 22. PMID 28943117

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study conducted at the University of Pennsylvania School of Dental Medicine. 240 South 40th Street, Robert Schattner Center, Philadelphia, PA 19104. Recruitment was from normal volunteers.
Period: Overall Study
Arm/Group | One Spray CTY-5339-A, Then One Spray CTY-5339-CB | 2 Sprays CTY-5339-A, Then 1 Spray CTY-5339-CB +1 Spray Placebo | One Spray of CTY-5339-CB, Then One Spray CTY-5339-A | 1 Spray CTY-5339-CB +1 Spray Placebo, Then 2 Sprays CTY-5339-A
Started | 10 | 10 | 10 | 10
Completed | 10 | 10 | 10 | 10
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- One Spray of CTY-5339-CB, Then One Spray CTY-5339-A: Two sprays of CTY-5339-A Anesthetic Spray (14.0% benzocaine and 2.0% tetracaine HCl) tested over a 60 minute session, followed by a 4-14 day washout period, followed by a single spray of CTY-5339-CB Anesthetic Spray (14.0% benzocaine) and a single spray of vehicle control (CTY-5339-P) (sprayed outside the circumscribed area to avoid dilution of active drug) tested over a 60 minute session.
- Total: Total of all reporting groups
Arm/Group | One Spray CTY-5339-A, Then One Spray CTY-5339-CB | 2 Sprays CTY-5339-A, Then 1 Spray CTY-5339-CB +1 Spray Placebo | One Spray of CTY-5339-CB, Then One Spray CTY-5339-A | 1 Spray CTY-5339-CB +1 Spray Placebo, Then 2 Sprays CTY-5339-A | Total
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 10 | 10 | 40
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.6 (9.0) | 25.0 (1.8) | 26.4 (2.8) | 27.6 (6.4) | 26.9 (5.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 4 | 9 | 25
  Male | 4 | 4 | 6 | 1 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 10 | 10 | 10 | 10 | 40
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 1
  Asian | 2 | 2 | 6 | 1 | 11
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 0 | 2 | 4
  White | 6 | 6 | 3 | 7 | 22
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 10 | 10 | 40
Weight (lbs) [Mean (Standard Deviation); unit: lbs] | 163.6 (38.3) | 153.6 (31.8) | 151.4 (33.7) | 144.5 (18.0) | 153.3 (30.9)
Height (inches) [Mean (Standard Deviation); unit: inches] | 66.7 (3.4) | 67.1 (2.6) | 68.3 (2.3) | 67.0 (2.9) | 67.3 (2.8)

OUTCOME MEASURES:

1. Primary Outcome: Duration of Anesthesia as Measured by Pin Prick Test (PPT) for One Spray CTY-5339-A Compared to One Spray CTY-5339-CB
Description: Evaluations were completed at 1-minute intervals for the first 5 minutes to capture onset of anesthesia. Starting at 5 minutes after drug administration, the PPT was done at 5 minute intervals up to the one hour time point. If there was no indication of anesthesia by 10 minutes, the subject was considered a treatment failure and the assessment of PPT was discontinued. In addition, once onset of anesthesia had occurred, if there was no longer any anesthesia at two consecutive evaluation time points from 10 minutes onward, the assessment of PPT was discontinued.
  The PPT was assessed using a 90-mm, 26-gauge pencil-point spinal needle. At screening, 3 pin pricks were performed on each cheek. Pin pricks were assessed using a 0 (no pain) to 10 (severe pain) Numerical Rating Scale (NRS). In order to be eligible for the study, for each cheek, subjects must have had a minimum score of "3" for the last 2 pin pricks, and one of those scores had to be "4" or higher.
Time Frame: Change in pain assessment from baseline (time of application) up to one hour post-application
Population: Modified Intent-to-Treat (mITT) population: all randomized subjects who, as documented prior to the breaking of the study blind: (1) met all the inclusion and exclusion criteria and; (2) either completed the two 60 minute test sessions or returned to baseline values in all evaluation tests.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | One Spray CTY-5339-A | One Spray CTY-5339-CB
Number analyzed (Participants) | 18 | 18
minutes | 17.9 (12.9) | 16.4 (14.8)
Statistical Analysis 1: Comparison: One Spray CTY-5339-A vs One Spray CTY-5339-CB; Test type: Superiority; p = 0.322, ANOVA; Mean Difference (Final Values) = 2.8, 95% CI 2-sided [-3.06 to 8.69], Standard Error of Mean 2.74 — Least squares mean (marginal mean)

2. Primary Outcome: Duration of Anesthesia as Measured by Heat Sensation Threshold (QST Heat) for One Spray CTY-5339-A Compared to One Spray CTY-5339-CB
Description: Starting at 5 minutes after drug administration, the QST was done at 5 minute intervals up to the one hour time point. If there was no indication of anesthesia by 10 minutes, the subject was considered a treatment failure and the assessment of PPT was discontinued. In addition, once onset of anesthesia had occurred, if there was no longer any anesthesia at two consecutive evaluation time points from 10 minutes onward, the assessment of QST was discontinued.
  The heat stimuli were delivered in 3 repetitions, with inter-stimulus intervals of 30s. The basal thermode temperature was set at a comfortable 35ºC. The rate at which the thermode heated up was set at 0.5ºC/s, while the rate at which it cooled down was set at 8ºC/s. The maximum thermode temperature was set at 51ºC. Heat sensation threshold was defined as the temperature at which the subjects first felt tingling, warmth, heat, or pain.
Time Frame: Change in temperature from baseline (time of application) up to one hour post-application
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | One Spray CTY-5339-A | One Spray CTY-5339-CB
Number analyzed (Participants) | 19 | 18
minutes | 44.6 (17.8) | 51.1 (12.9)
Statistical Analysis 1: Comparison: One Spray CTY-5339-A vs One Spray CTY-5339-CB; Test type: Superiority; p = 0.134, ANOVA; Mean Difference (Final Values) = -8.7, 95% CI 2-sided [-20.38 to 2.99], Standard Error of Mean 5.48 — Least squares mean (marginal mean)

3. Secondary Outcome: Duration of Anesthesia as Measured by Pin Prick Test (PPT) for Two Sprays CTY-5339-A Compared to One Spray CTY-5339-CB in Combination With One Spray CTY-5339-P (Placebo)
Description: Assessments will be made over a period of one hour, with assessments at 1 minute intervals for the first 5 minutes and then every 5 minutes after that. Duration of effect was defined as the time (in minutes) from onset to treatment failure (i.e., for PPT, an assessment of "Same/More" pain, and for QST, the average heat temperature was greater than the average heat temperature at Baseline (non-treated cheek), up to the 60-minute time point (at two consecutive time points).
Time Frame: Time of application up to one hour post-application
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Minutes
Groups:
- One Spray CTY-5339-CB in Combination With One Spray CTY-5339-P: A single spray of CTY-5339-CB in a metered spray bottle with ≈200 uL total spray volume, containing the active ingredient: 14.0% Benzocaine (USP = 28 mg). This was administered in combination with a single spray of CTY-5339-P (acting as vehicle control placebo with no active ingredient) in a metered spray bottle with ≈200 uL total spray volume. This combination was used to maintain double-blind conditions. The vehicle control was sprayed outside the circumscribed area to avoid dilution of active drug.
Arm/Group | Two Sprays CTY-5339-A | One Spray CTY-5339-CB in Combination With One Spray CTY-5339-P
Number analyzed (Participants) | 18 | 17
Minutes | 17.3 (17.0) | 13.5 (14.7)
Statistical Analysis 1: Comparison: Two Sprays CTY-5339-A vs One Spray CTY-5339-CB in Combination With One Spray CTY-5339-P; Test type: Superiority; p = 0.442, ANOVA; Mean Difference (Final Values) = 4.1, 95% CI 2-sided [-6.48 to 14.62], Standard Error of Mean 4.92 — Least squares mean (marginal mean)

4. Secondary Outcome: Duration of Anesthesia as Measured by QST Heat for Two Sprays CTY-5339-A Compared to One Spray CTY-5339-CB in Combination With One Spray CTY-5339-P (Placebo)
Description: as for outcome 3
Time Frame: Time of application up to one hour post-application
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Two Sprays CTY-5339-A | One Spray CTY-5339-CB in Combination With One Spray CTY-5339-P
Number analyzed (Participants) | 19 | 20
minutes | 46.8 (17.3) | 38.9 (20.3)
Statistical Analysis 1: Comparison: Two Sprays CTY-5339-A vs One Spray CTY-5339-CB in Combination With One Spray CTY-5339-P; Test type: Superiority; p = 0.172, ANOVA; Mean Difference (Final Values) = 6.8, 95% CI 2-sided [-3.27 to 16.90], Standard Error of Mean 4.78 — Least squares mean (marginal mean)

5. Secondary Outcome: Duration of Anesthesia as Measured by PPT for One Spray CTY-5339-A Compared to Two Sprays CTY-5339-A
Description: Assessments will be made over a period of one hour, with assessments at 1 minute intervals for the first 5 minutes and then every 5 minutes after that.
Time Frame: Time of application up to one hour post-application
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | One Spray CTY-5339-A | Two Sprays CTY-5339-A
Number analyzed (Participants) | 18 | 18
minutes | 17.9 (12.9) | 17.3 (17.0)

6. Secondary Outcome: Duration of Anesthesia as Measured by QST Heat for One Spray CTY-5339-A Compared to Two Sprays CTY-5339-A
Description: as for outcome 5
Time Frame: Time of application up to one hour post-application
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | One Spray CTY-5339-A | Two Sprays CTY-5339-A
Number analyzed (Participants) | 19 | 19
minutes | 44.6 (17.8) | 46.8 (17.3)

7. Secondary Outcome: Onset of Anesthesia for PPT
Description: as for outcome 5
Time Frame: Time of application up to one hour post-application
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | One Spray CTY-5339-A | Two Sprays CTY-5339-A | One Spray CTY-5339-CB | One Spray CTY-5339-CB in Combination With One Spray CTY-5339-P
Number analyzed (Participants) | 18 | 18 | 18 | 17
Minutes | 1.2 (0.4) | 1.5 (0.9) | 1.7 (2.1) | 1.7 (1.3)

8. Secondary Outcome: Onset of Anesthesia for QST Heat
Description: as for outcome 5
Time Frame: Time of application up to one hour post-application
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Minutes
Groups:
- CTY-5339-CB 1 Spray + Placebo 1 Spray: Benzocaine and Placebo; 14.0% Benzocaine, USP = 28 mg; 200 uL and one spray Vehicle control (no active ingredient); 200 uL
Arm/Group | One Spray CTY-5339-A | Two Sprays CTY-5339-A | One Spray CTY-5339-CB | CTY-5339-CB 1 Spray + Placebo 1 Spray
Number analyzed (Participants) | 19 | 19 | 18 | 20
Minutes | 3.1 (3.3) | 1.9 (1.4) | 1.7 (1.3) | 4.2 (5.2)

9. Secondary Outcome: Percentage of Responders for PPT at Each Time Point
Description: as for outcome 5
Time Frame: Time of application up to one hour post-application
Population: Some treatment response data was missing or lost or an invalid value was recorded
Measure: Count of Participants; unit: Participants
Arm/Group | One Spray CTY-5339-A | Two Sprays CTY-5339-A | One Spray CTY-5339-CB | One Spray CTY-5339-CB in Combination With One Spray CTY-5339-P
Number analyzed (Participants) | 20 | 20 | 20 | 20
Participants
  Responded to treatment at the 1 minute time point: number analyzed (Participants) | 20 | 19 | 20 | 19
  Responded to treatment at the 1 minute time point | 12 | 12 | 14 | 10
  Responded to treatment at the 2 minute time point: number analyzed (Participants) | 20 | 19 | 20 | 19
  Responded to treatment at the 2 minute time point | 13 | 9 | 14 | 13
  Responded to treatment at the 3 minute time point: number analyzed (Participants) | 20 | 19 | 20 | 19
  Responded to treatment at the 3 minute time point | 12 | 11 | 12 | 10
  Responded to treatment at the 4 minute time point: number analyzed (Participants) | 20 | 19 | 20 | 19
  Responded to treatment at the 4 minute time point | 12 | 12 | 8 | 8
  Responded to treatment at the 5 minute time point: number analyzed (Participants) | 20 | 19 | 20 | 19
  Responded to treatment at the 5 minute time point | 10 | 7 | 7 | 9
  Responded to treatment at the 10 minute time point: number analyzed (Participants) | 20 | 19 | 20 | 19
  Responded to treatment at the 10 minute time point | 5 | 6 | 8 | 6
  Responded to treatment at the 15 minute time point: number analyzed (Participants) | 20 | 20 | 20 | 19
  Responded to treatment at the 15 minute time point | 8 | 5 | 6 | 4
  Responded to treatment at the 20 minute time point | 4 | 6 | 4 | 2
  Responded to treatment at the 25 minute time point | 3 | 5 | 4 | 1
  Responded to treatment at the 30 minute time point | 3 | 6 | 2 | 2
  Responded to treatment at the 35 minute time point | 1 | 3 | 1 | 1
  Responded to treatment at the 40 minute time point | 1 | 0 | 0 | 1
  Responded to treatment at the 45 minute time point | 0 | 1 | 1 | 1
  Responded to treatment at the 50 minute time point | 0 | 1 | 0 | 1
  Responded to treatment at the 55 minute time point | 0 | 0 | 1 | 1
  Responded to treatment at the 60 minute time point | 0 | 0 | 0 | 1

10. Secondary Outcome: Percentage of Responders for QST Heat at Each Time Point
Description: as for outcome 5
Time Frame: Time of application up to one hour post-application
Population: A baseline measure was lost/missing for one treatment so the response could not be calculated.
Measure: Count of Participants; unit: Participants
Arm/Group | One Spray CTY-5339-A | Two Sprays CTY-5339-A | One Spray CTY-5339-CB | One Spray CTY-5339-CB in Combination With One Spray CTY-5339-P
Number analyzed (Participants) | 20 | 19 | 20 | 20
Participants
  Responded to treatment at the 5 minute time point | 16 | 18 | 18 | 15
  Responded to treatment at the 10 minute time point | 17 | 17 | 17 | 13
  Responded to treatment at the 15 minute time point | 15 | 17 | 18 | 15
  Responded to treatment at the 20 minute time point | 17 | 15 | 17 | 14
  Responded to treatment at the 25 minute time point | 15 | 15 | 15 | 14
  Responded to treatment at the 30 minute time point | 14 | 14 | 14 | 13
  Responded to treatment at the 35 minute time point | 13 | 12 | 17 | 12
  Responded to treatment at the 40 minute time point | 12 | 11 | 16 | 12
  Responded to treatment at the 45 minute time point | 13 | 11 | 12 | 11
  Responded to treatment at the 50 minute time point: number analyzed (Participants) | 20 | 19 | 19 | 20
  Responded to treatment at the 50 minute time point | 9 | 12 | 10 | 10
  Responded to treatment at the 55 minute time point: number analyzed (Participants) | 20 | 19 | 19 | 20
  Responded to treatment at the 55 minute time point | 9 | 11 | 9 | 9
  Responded to treatment at the 60 minute time point: number analyzed (Participants) | 20 | 19 | 19 | 20
  Responded to treatment at the 60 minute time point | 10 | 11 | 10 | 8

ADVERSE EVENTS:
Time Frame: Adverse event data collected during and for one hour post testing.
Groups:
- CTY-5339-A 1 Spray: Benzocaine and Tetracaine 14.0% Benzocaine, USP = 28 mg 2.0% Tetracaine Hydrochloride, USP = 4 mg
  Benzocaine and Tetracaine: A single application 1 spray of a combination of benzocaine 14% and tetracaine 2% with a total dose of benzocaine 28 mg and tetracaine 2 mg per spray.
- CTY-5339-A 2 Sprays: Benzocaine and Tetracaine 14.0% Benzocaine, USP = 56 mg 2.0% Tetracaine Hydrochloride, USP = 8 mg
  Benzocaine and Tetracaine: A single application of 2 sprays of a combination of benzocaine 14% and tetracaine 2% with a total dose of benzocaine 28 mg and tetracaine 2 mg per spray.
- CTY-5339-CB 1 Spray: Benzocaine only 14.0% Benzocaine, USP = 28 mg
  Benzocaine only: Benzocaine 14% alone 200 uL (1 spray)
  A single application of 1 spray of benzocaine 14% with a total dose of benzocaine 28 mg.
- CTY-5339-CB 1 Spray + Placebo 1 Spray: Benzocaine and Placebo 14.0% Benzocaine, USP = 28 mg; 200 uL and one spray Vehicle control (no active ingredient); 200 uL
  A single application of 1 spray of benzocaine 14% and a single spray of placebo with a total dose of benzocaine 28 mg.
Arm/Group | CTY-5339-A 1 Spray | CTY-5339-A 2 Sprays | CTY-5339-CB 1 Spray | CTY-5339-CB 1 Spray + Placebo 1 Spray
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20 | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 1/20 | 0/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CTY-5339-A 1 Spray (N=20) | CTY-5339-A 2 Sprays (N=20) | CTY-5339-CB 1 Spray (N=20) | CTY-5339-CB 1 Spray + Placebo 1 Spray (N=20)
Feeling faint (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Dizziness; Mild Severity; Unrelated to study medication; Resolved, no sequelae

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-11-10): https://cdn.clinicaltrials.gov/large-docs/20/NCT02908620/Prot_SAP_000.pdf